CLINICAL TRIAL: NCT00264368
Title: Ganciclovir Pharmacokinetics in Patients Undergoing Continuous Renal Replacement Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCV-PRISMA
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Acute Renal Failure; Cytomegalovirus Infections; Multi Organ Failure
Keywords: Renal replacement therapy; CMV disease
MeSH Terms: conditions — Acute Kidney Injury; Cytomegalovirus Infections; Multiple Organ Failure | interventions — Ganciclovir

INTERVENTIONS:
Drug: intravenous (IV) ganciclovir

SUMMARY:
In order to optimize anti-cytomegalovirus (CMV) treatment with ganciclovir (GCV), in patients with multi organ failure treated with continuous renal replacement therapy (RRT), more information about ganciclovir pharmacokinetics in this setting is needed.

The primary objective is to describe the pharmacokinetics of ganciclovir in critically ill patients with acute renal failure treated with continuous renal replacement therapy, with a special emphasis on the extra-renal clearance and distribution volume.

Secondary objectives are to investigate if any co-factors, such as serum creatinine, weight, general hydration status, rest function of the native kidneys, etc. can help to describe the pharmacokinetics of GCV in these patients on continuous RRT as well as the relative influence of filtrations and dialysis on GCV elimination during different modalities of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of continuous RRT and GCV treatment
* 18 years of age or older.

Exclusion Criteria:

* Concomitant treatment with acyclovir or valacyclovir.
* Patient does not give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2005-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
comparing the total clearance with the RRT derived clearance of GCV
comparing the volume of distribution with historic controls of non Intensive Care Unit (ICU) patients

SECONDARY OUTCOMES:
comparing GCV plasma concentration and population model derived estimates of these concentrations when including different relevant clinical co-factors such as: weight, S-creatinine, CL-creatinine, hydration, albumin, rest function of native kidneys etc.
determine RRT derived GCV clearance during the different filtration/dialysis settings of the RRT machine

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, Ph.D., Study Director — University of Oslo School of Pharmacy; Anders Hartmann, MD, Ph.D., Principal Investigator — Rikshospitalet, Medical Department; Jan F Bugge, MD, Ph.D., Study Chair — Rikshospitalet, Department of Anaesthesiology
Locations (1):
- Rikshospitalet, Section of Nephrology, Oslo, Norway